CLINICAL TRIAL: NCT04437732
Title: 30 Day Trial Fitting of a New Bifocal Contact Lens
Brief Title: Apioc Presbyopic Contact Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lentechs, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: LEN-002
Record Dates: First submitted 2020-06-16; First posted 2020-06-18 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: Presbyopia; Refractive Errors
Keywords: contact lens; soft contact lens
MeSH Terms: conditions — Presbyopia; Refractive Errors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Apioc Lens (Other): All subjects will wear either the Apioc-P or Apioc-PT contact lens design
  Interventions: Device: Apioc-P and Apioc-PT Contact Lens Design

INTERVENTIONS:
Device: Apioc-P and Apioc-PT Contact Lens Design — Novel soft contact lens design

SUMMARY:
In this study, you will wear an invesetigational contact lens, Apioc-P or Apioc-PT, the way you wear your current contact lenses for approximately one month (no more than 35 days).

DETAILED DESCRIPTION:
Apioc-P and Apioc-PT is an investigational contact lens, which means it has not been approved by the U.S. Food and Drug Administration (FDA), although the contact lens material, called Definitive 74, is already approved and marketed for contact lenses that are similar to Apioc-P and Apioc-PT. In this study, participants will wear an Apioc-P and Apioc-PT contact lens the way they wear their current contact lenses for approximately one month (no more than 35 days).

Participation in this study will include a minimum of four study visits. The first will last up to 90 minutes, the second will last up to 45 minutes, the third will last up to 45 minutes, and the final visit will be up to 90 minutes. If the lens does not appear to be fitting properly at the second visit, then another lens will be ordered for participants and they will be asked to return for an additional visit for up to 45 minutes. Up to 60 subjects will participate in this study.

ELIGIBILITY:
Inclusion Criteria:

1. The subject must provide written informed consent.
2. The subject must appear willing and able to adhere to the instructions set forth in this protocol.
3. At least 40 years of age and no more than 70 years of age.
4. ≤ 4.00 D of corneal astigmatism.
5. ≤ 4.00 D of refractive astigmatism.
6. Refractive error range +20.00 DS to -20.00 DS
7. Keratometry readings within 40 to 50D.
8. Clear, healthy corneas with no irregular astigmatism.
9. Normal, healthy conjunctiva in both eyes.
10. Free of active ocular disease. Refractive error and presbyopia are permitted.
11. Be a current or former (within the last 12 months) contact lens wearer.
12. Best-corrected near and distance visual acuity better than or equal to 20/25.

Exclusion Criteria:

1. Irregular corneal astigmatism.
2. Corneal scarring unless off line-of-site and well healed.
3. Pinguecula, pterygium, or other conjunctival thickness abnormalities that would interfere with soft contact lens wear.
4. Recent use of any ocular pharmaceutical treatments, including daily artificial tears, in the two weeks prior to the examination. Use of artificial tears less than 3 times per week is permitted.
5. Systemic disease that would interfere with contact lens wear.
6. Currently pregnant or lactating (by self-report).
7. History of strabismus or eye movement disorder, including exophoria at near that is 4D or greater than at far, and a receded near point of convergence break that is 6 cm or greater.
8. Active allergies that may inhibit contact lens wear.
9. Upper eyelid margin at or above the superior limbus.
10. History of ocular or lid surgery.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2019-11-11 (Actual); Primary Completion 2021-06-09 (Actual); Study Completion 2021-06-09 (Actual)

PRIMARY OUTCOMES:
Visual Acuity | 30 days
  LogMAR visual acuity

SECONDARY OUTCOMES:
Comfort | 30 days
  Contact Lens Dry Eye Questionnaire-8, scale range 0 minimum (better outcome) to 38 maximum (worse outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Thomas G Quinn, OD, MS, FAAO, Principal Investigator — Drs. Quinn, Foster & Associates; Jason R Miller, OD, MBA, Principal Investigator — Eyecare Professionals of Powell
Locations (2):
- United States (2):
  - Quinn Foster & Associates, Athens, Ohio
  - EyeCare Professionals of Powell, Powell, Ohio

IPD SHARING:
Plan to Share IPD: No